CLINICAL TRIAL: NCT05755659
Title: Clinical on the Safety and Effectiveness of Fosaprepitant Dimeglumine for Injection in the Prevention of Nausea and Vomiting Caused by Tumor Chemotherapy Drugs.
Brief Title: Clinical on the Safety and Efficacy of Fosaprepitant Dimeglumine for Injection in the Prevention of CINV.
Acronym: COSEFDIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TQXB-SQ001
Record Dates: First submitted 2023-01-10; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — fosaprepitant; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor chemotherapy patients (Experimental): To evaluate the safety of Fosaprepitant Dimeglumine for injection in the prevention of nausea and vomiting caused by tumor chemotherapy drugs
  Interventions: Drug: Fosaprepitant Dimeglumine for Injection

INTERVENTIONS:
Drug: Fosaprepitant Dimeglumine for Injection — The specification of Fosaprepitant Dimeglumine for injection is 150 mg, and the usage and dosage is: when preventing nausea and vomiting caused by HEC, this product is used in combination with dexamethasone and 5-HT3 antagonist. The dosage of Fosaprepitant Dimeglumine for injection is 150 mg, and the infusion time is 20-30 minutes. The intravenous infusion is completed 30 minutes before the beginning of chemotherapy on the first day.
  Other Names: ShanQi®️

SUMMARY:
To evaluate the safety of Fosaprepitant Dimeglumine Injection for the prevention of nausea and vomiting caused by tumor chemotherapy drugs, analyze the characteristics of the applicable population and clinical medication of Fosaprepitant Dimeglumine, evaluate the risk factors that may affect the efficacy of drug use, and compare the clinical benefits of different drug use modes.

DETAILED DESCRIPTION:
This is a prospective, one arm, open, non-interference, multi center, observational, real world clinical study.

Study drug: Fosaprepitant Dimeglumine for injection. White or almost white lump or powder, containing 150mg (calculated as C23H22F7N4O6P). This product is a NK-1 receptor antagonist, which is administered jointly with other antiemetic drugs. It is suitable for adult patients to prevent acute and delayed nausea and vomiting during the initial and repeated treatment of highly emetic chemotherapy drugs (HEC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with nausea and vomiting caused by chemotherapy
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Hypersensitive to any component in this product
* Patients taking pimozide, terfenadine, astemizole and cisapride

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Safety of Fosaprepitant Dimeglumine | 7 day
  Safety evaluation: observe the known adverse reactions (including those found in preclinical studies, clinical studies, previous routine monitoring, and those in the same product of aspirin) and whether there are new adverse reactions, and observe the incidence and occurrence of these adverse reactions (occurrence characteristics, severity, risk factors), At the same time, we should pay attention to the occurrence of adverse reactions of drugs used in special groups (pregnant women, children, the elderly, patients with liver and kidney dysfunction), and the safety of different chemotherapy schemes.
Effectiveness of Fosaprepitant Dimeglumine | 7 day
  Efficacy evaluation: complete control rate (CR), that is, the proportion of patients without vomiting and without remedial drugs; Including acute CR (0-24h) and delayed vomiting CR (25-120h). To evaluate the applicable population characteristics and clinical medication characteristics of fosapitam, observe the efficacy of fosapitam in different chemotherapy schemes, tumor types and different dosage schemes, preliminarily analyze the risk factors affecting the efficacy of fosapitam, and compare the clinical benefits of different medication modes.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, Study Chair — Digestive surgery
Locations (1):
- The First Affiliated Hospital of Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No